CLINICAL TRIAL: NCT05820360
Title: Cognitive Model for Behavioral Interventions (CoMBI) as a Personalized Behavioral Intervention for Patients With Serious Mental Illness
Brief Title: Cognitive Model for Behavioral Interventions as a Personalized Intervention for Patients With Serious Mental Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Saskia Bollen, Principal Investigator, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoMBI-SMI
Record Dates: First submitted 2023-04-07; First posted 2023-04-19 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Model Description:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with Serious Mental Illness (Experimental): The target groups are adult (18 to 65 years) and elderly (over 65 years) patients with a Serious Mental Illness. Inclusion criteria: presence of SMI and behavioral problems, willingness and ability to participate in this research.
  Interventions: Behavioral: CoMBI-SMI

INTERVENTIONS:
Behavioral: CoMBI-SMI — The first step is analysis of the behavioral problem because the core need is insufficiently compensated by the current environment or counteracted by the behavior of people within that environment. Step 2 is to choose the right core need based on this analysis. CoMBI-SMI describes the patient's self-image, the image of others, the triggering events and the problematic behavior of the patient based on personality disorders as classified by the Diagnostical and Statistical Manual of Mental Disorders. Step 3 is to choose the nursing intervention that is easily deployable so that Healthcare providers can identify the underlying core need and reduce the behavioral problems and burden on the healthcare providers. The fourth and final step is to draw up a CoMBI plan. The CoMBI-SMI is a cyclical process where it is important that the entire team is aligned with the patient's behavioral approach. Interventions are carried out by the entire team and evaluated after an agreed period of time.

SUMMARY:
The aim of this clinical study is to investigate whether CoMBI-SMI helps to reduce behavioral problems and psychiatric complaints in Serious Mental Illness (SMI) populations complaints and to reduce the burden on informal caregivers. It will also be examined whether there is an improvement in the quality of life of the participants. Participants are asked to complete two questionnaires. Then the participants receive treatment as is normally given in a clinical department. In particular, the caregivers will be asked to observe the behavior of the participants using a questionnaire and to follow a CoMBI-training to better tailor the treatment to the core needs of the participants. Comparisons will be made within the participant group because measurements take place before and after the procedure.

DETAILED DESCRIPTION:
In this study, the effectiveness of a treatment protocol for a personalized approach to behavioral problems, based on the core needs of patients based on their specific personality traits will be investigated. Patients will be recruited from clinical departments of (top) specialist mental health care institutions. Both adult (18-64 years old) and older adults (≥ 65 years) patients with SMI will be included in this study. Primary outcome measures are the Neuropsychiatric Inventory-Questionnaire (NPI-Q) and Brief Symptom Inventory (BSI). Secondary outcome measures are the burden of care for the team and the patient's quality of life, measured with the NPI-Q and Mental Health Quality of life (MHQoL-7D), respectively. Furthermore, predictive factors are mapped for the primary and secondary outcome measures. The gathered NPI-Q data will then be used for a validation study, where the construct validity, internal consistency and inter-rater reliability of the NPI-Q in an SMI population will be assessed.

Individual or group psychotherapy for SMI is not always possible because several patients are unwilling or unable to accept such treatment. Mediation therapy is an alternative, in which interventions are used via a team of professionals to bring about behavioral change in the patient. Unfortunately, there are only a few guidelines and protocols available in the field of mediation therapy. Therefore, the aim of this study will be the development of CoMBI-SMI for the SMI-population. CoMBI-SMI is a combination of cognitive behavioral therapy based upon Beck's cognitive model of personality disorders and nursing interventions from the Nursing Interventions Classification. Triggers from the environment may create a behavioral problem that is maintained by its consequences. The behavioral problems are first identified by the team. Based on this analysis, a core need is selected from the CoMBI-SMI protocol and the associated nursing interventions are selected. This is described in a CoMBI-plan and evaluated cyclically.

Healthcare providers of the departments will be trained in CoMBI-SMI. The training will consist of an online theoretical part about the model followed by a Meet-The-Expert meeting (MTE), where healthcare providers can ask questions about the theoretical part and where CoMBI-SMI will be practiced on the basis of case studies. Quality criteria are linked to the online training, wherein the theoretical part is tested by means of case studies.

According to a stepped wedge design cross-overtime from condition A to CoMBI-SMI varies across participating teams. Condition A is treatment as usual (TAU) with measurements each 4 weeks and the effect is measured by the NPI-Q, BSI and the MHQoL-7D. To properly identify the core needs for the CoMBI-SMI approach, the personality questionnaires Personality Inventory for Diagnostic and Statistical Manual of Mental Disorders edition 5 (PID-5-Brief form+Modified) and the Level of Personality Functioning-scale brief 2.0 (LPFS-Brief form 2.0) will be used. Then, the CoMBI training takes place and CoMBI-SMI is performed with also measurements each 4 weeks and the effect is measured with the same outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* psychogeriatric inpatients aged 18+
* presence of SMI and behavioral problems
* willingness and ability to participate in this study.

Exclusion Criteria:

* behavioral problems caused by delirium
* current substance-related disorder
* treatment in forensic psychiatry at the time of study
* manic phase
* florid psychosis
* when the behavioral problems arise directly from acquired brain injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory - Questionnaire (NPI-Q) | Before the start of TAU, before the CoMBI-SMI training and after 4 weeks of CoMBI-SMI-training
  The NPI-Q was developed and validated in 2000 and translated into Dutch in 2002. The NPI-Q contains 12 domains that can be used to map neuropsychiatric symptoms. These domains are: delusions; hallucinations; agitation/aggression; depression/dysphoria; fear; euphoria / elation; apathy/indifference; disinhibited behavior; irritability/lability; aimless repetitive behavior; night restlessness/sleep disorder; appetite/eating behavior change. The questionnaire is completed by the patient's caregiver and charts whether a particular symptom is present or not, how severe this symptom is (on a three-point scale) if present, and how severe the emotional burden of this symptom is for the caregiver (on a six-point scale). The test-retest correlation of the NPI-Q for symptom severity is 0.80 and for emotional burden is 0.94. The convergent validity, compared to the NPI, is 0.91 for symptom severity and 0.92 for emotional burden.
Brief Symptom Inventory (BSI) | Before the start of TAU, before the CoMBI-SMI training and after 4 weeks of CoMBI-SMI-training
  The Brief Symptom Inventory (BSI) is a multidimensional complaints list that shows the extent to which the patient suffered from psychological and/or physical symptoms during the past period. This test also gives a score for the total number of complaints, the total symptoms present and the severity of the symptoms present. The test consists of 53 items scored from "not at all = 0" to "very much = 4". There are 9 subscales: Somatic complaints; Cognitive problems; Interpersonal sensitivity; Depressed mood; Fear; Hostility; Phobic fear; Paranoid thoughts; Psychoticism. The test is sensitive to therapy influences. The BSI is a sufficiently reliable and valid test. The test is standardized for the Dutch language area with the norm groups men vs. women and general population vs. patients. The currently available norm groups were established in 2011.

SECONDARY OUTCOMES:
Mental Health Quality of Life (MHQoL-7D) | Before the start of TAU, before the CoMBI-SMI training and after 4 weeks of CoMBI-SMI-training
  The Mental Health Quality of Life (MHQoL-7D) measures the quality of life in people with mental health problems. The MHQoL-7D is a standardized instrument consisting of two parts: a descriptive section, the MHQoL-7D, and a visual analog scale. The MHQoL-7D consists of seven questions covering seven dimensions, each with four response levels ranging from very satisfied to very dissatisfied: self-esteem, independence, mood, relationships, daily activities, physical health, and future. The total score can range from 0 to 21; the higher the score, the better the quality of life. The MHQoL visual analog scale measures the respondent's general psychological well-being on a horizontal scale ranging from zero, 'only imaginable psychological well-being' to ten, 'best imaginable psychological well-being'.

OTHER OUTCOMES:
Personality Inventory for Diagnostic and Statistical Manual of Mental Disorders edition 5 (PID-5-BF+Modified) | Once before the start of the CoMBI-SMI training.
  The Personality Inventory for Diagnostic and Statistical Manual of Mental Disorders edition 5 is a 220-item self-report list of five domains (Negative Affectivity, Detachment, Antagonism, Disinhibition and Psychoticism) and the 25 associated facets of Criterion B measured from the Alternative Personality Disorder Model. The instrument can be used as a reliable screening measure for dimensional maladaptive personality traits. From the longer version PID-5-dutch version it is possible to use the shorter version, the PID-5-Brief form+Modified. The proposed study uses the shortened self-report version and informant version of the derived Dutch version, the PID-5-Brief form+Modified. This version consists of 36 self-report items (all part of the original PID-5) and covers a combination of the five Diagnostic and Statistical Manual of Mental disorders edition 5 domains and the Internation Classification of diseases edition 11 personality trait domain Anankastic, resulting in six domains.
Level of Personality Functioning-scale brief form 2.0 | Once before the start of the CoMBI-SMI training.
  The LPFS-brief form 2.0 measures the level of personality functioning as described in the Diagnostic and Statistical Manual of mental Disorders with items for the four domains of personality functioning (identity, self-direction, empathy and intimacy) (Rossi et al., 2019). There are three items for each of the four domains, resulting in 12 items.The items measure the four domains of Criterion A to determine the severity of the personality disorder. It is a self-report questionnaire originally developed in Dutch. There is also an informant version. A preliminary study in a clinical sample including younger adults found evidence for a factor structure of two overarching factors, self and interpersonal functioning, that showed relevant associations with different severity measures. In addition, the LPFS-Brief form 2.0 has been shown to have good convergent validity in older adults in a clinical sample.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Bollen, Principal Investigator — Vrije Universiteit Brussel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Kat MG, de Jonghe JF, Aalten P, Kalisvaart CJ, Droes RM, Verhey FR. [Neuropsychiatric symptoms of dementia: psychometric aspects of the Dutch Neuropsychiatric Inventory (NPI)]. Tijdschr Gerontol Geriatr. 2002 Sep;33(4):150-5. Dutch. PMID 12378786
- [Background] de Beurs E, den Hollander-Gijsman ME, van Rood YR, van der Wee NJ, Giltay EJ, van Noorden MS, van der Lem R, van Fenema E, Zitman FG. Routine outcome monitoring in the Netherlands: practical experiences with a web-based strategy for the assessment of treatment outcome in clinical practice. Clin Psychol Psychother. 2011 Jan-Feb;18(1):1-12. doi: 10.1002/cpp.696. PMID 20238371
- [Background] van Krugten FCW, Busschbach JJV, Versteegh MM, Hakkaart-van Roijen L, Brouwer WBF. The Mental Health Quality of Life Questionnaire (MHQoL): development and first psychometric evaluation of a new measure to assess quality of life in people with mental health problems. Qual Life Res. 2022 Feb;31(2):633-643. doi: 10.1007/s11136-021-02935-w. Epub 2021 Jul 9. PMID 34241821
- [Background] Krueger RF, Derringer J, Markon KE, Watson D, Skodol AE. Initial construction of a maladaptive personality trait model and inventory for DSM-5. Psychol Med. 2012 Sep;42(9):1879-90. doi: 10.1017/S0033291711002674. Epub 2011 Dec 8. PMID 22153017
- [Background] Anderson JL, Sellbom M. Evaluating the DSM-5 Section III personality disorder impairment criteria. Personal Disord. 2018 Jan;9(1):51-61. doi: 10.1037/per0000217. Epub 2016 Sep 12. PMID 27618341
- [Background] Osterloh JWSA, Videler AC, Rossi GMP, van Alphen SPJ. [Cognitive model for behavioural interventions for personality disorders in older adults: a nursing approach]. Tijdschr Gerontol Geriatr. 2018 Oct;49(5):210-212. doi: 10.1007/s12439-018-0256-6. Epub 2018 Jul 31. Dutch. PMID 30066308
- [Background] Bach B, Hutsebaut J. Level of Personality Functioning Scale-Brief Form 2.0: Utility in Capturing Personality Problems in Psychiatric Outpatients and Incarcerated Addicts. J Pers Assess. 2018 Nov-Dec;100(6):660-670. doi: 10.1080/00223891.2018.1428984. Epub 2018 Mar 1. PMID 29494782
- [Background] Rossi, G., Debast, I., Berghuis, H., Ingenhoven, T. J. M., van der Heijden, P., & Morey, L. (2019).Nederlandstalige vertaling van de niveaus van persoonlijkheidsfunctioneren zelfrapportage schaal (Level ofPersonality Functioning Scale-Self Report; LPFS-SR).